CLINICAL TRIAL: NCT00687856
Title: Identifying and Facilitating Ventricular Recovery on Mechanical Support
Acronym: RECOVER
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 585; R01HL086918 (NIH)
Record Dates: First submitted 2008-05-29; First posted 2008-06-02 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2023-10-16 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure
Keywords: Left Ventricular Assist Device
MeSH Terms: conditions — Heart Failure | interventions — Caves

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- LVAD Recipients: Participants who have had or are about to have a left ventricular assist device (LVAD) implanted
  Interventions: Procedure: Echocardiogram (echo)

INTERVENTIONS:
Procedure: Echocardiogram (echo) — Participants will undergo a series of echoes to determine if they are eligible to be weaned from LVAD support. Each echo exam will involve the use of an ultrasound probe on the chest of participants to assess the pumping ability of their hearts.

SUMMARY:
Heart failure is a progressive disorder in which the weakened heart is not able to efficiently pump blood throughout the body. When the body's cells do not receive enough blood, this can result in fatigue, shortness of breath, and difficulty carrying out daily activities. The left ventricular assist device (LVAD) is a device that is used to provide mechanical circulatory support to patients with end-stage heart failure who are awaiting heart transplants. Although LVAD support helps maintain the pumping ability of the heart and dramatically improves heart failure symptoms, the quality of life with LVAD support is far from ideal. It has been shown that LVAD support in selected patients may restore the failing heart enough to eliminate the need for heart transplant, but more information is needed to assess heart recovery and to guide weaning of LVAD support. Using data collected from patients who have undergone LVAD implantation, this study will attempt to better assess heart recovery and to generate criteria for identifying patients eligible for the removal of LVAD support.

DETAILED DESCRIPTION:
It is estimated that approximately 5 million people in the United States have heart failure, with more than 500,000 new cases diagnosed each year. Heart failure is a disorder that develops over many years and can be attributed to a number of conditions, including heart attack, coronary artery disease, diabetes, high blood pressure, or congenital heart defects. Although there are many treatment options for heart failure, people with end-stage heart failure may benefit most from a heart transplant. However, the number of donor organs available remains limited, making alternative treatments for people with end-stage heart failure imperative. LVAD support, which has traditionally been used as a bridge to transplant, may also provide an alternative life-saving measure for patients with advanced end-stage heart failure. The mechanical circulatory support provided by LVAD may allow the left side of the heart to rest and recover enough so that removal of the device is possible and a heart transplant is no longer needed, at least temporarily. However, more research in this area is needed. Using data collected from patients who have undergone LVAD implantation, this study will attempt to better assess heart recovery and to generate criteria for identifying patients eligible for the removal of LVAD support.

Participation in this study will last up to 3 years. First, 3 months before LVAD implantation, participants' medical records, including their medical history, medical therapy, and cardiac testing, will be obtained. Next, participants will undergo a weaning echocardiogram (echo) 1 month after LVAD implantation and, if necessary, monthly for 2 more months.During the weaning echoes, participants will have their LVAD settings adjusted, condition monitored, and additional data concerning their status collected. Before each echo, participants will also undergo a blood draw to determine how much blood thinner they will receive, if necessary.

12cc of blood will be collected up to 30 days prior to the VAD implant to look at gene expression and proteins expressed in your white blood cells and blood serum.

During the surgery, a small piece of tissue, ranging in the size from 1/4 inch cubed to 1 inch cubed will be removed from the heart tissue. The surgeon removes the heart tissue as part of the normal surgical process, so that the surgeon can implant the VAD. Approximately half of the tissue will then be stored for research purposes.

2-6 weeks after surgery a second blood draw of 12cc will be drawn again to look at the gene expression and proteins expressed in the patient's white blood cells and blood serum.

Participants who are not eligible to be weaned from LVAD support after the three weaning echoes will continue to be monitored every 6 months for up to 3 years or until the device is removed. Participants who are eligible to have the LVAD removed will undergo another echo after they have recovered from the surgery and are no longer taking any intravenous medications to help the heart. Data from any routine follow-up echoes will also be collected from these participants every 6 months until study completion at Year 3.

If the patient's heart recovers and the LVAD is removed, we are interested in removing a second piece of heart tissue that would otherwise be discarded at the time of removal of the LVAD.

ELIGIBILITY:
Inclusion Criteria:

* Eligible to receive an LVAD or biventricular assist device (BIVAD) for clinical indications.

Exclusion Criteria:

* Refuses LVAD support
* Requires right ventricular assist device (RVAD) placement alone
* In atrial fibrillation with a ventricular response of greater than 120 beats per minute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include participants who have undergone or are about to undergo LVAD implantation at one of the three participating clinical centers.
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2008-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Gorcsan, MD, Principal Investigator — UPMC University of Pittsburgh
Locations (5):
- United States (5):
  - University of Maryland, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - INTEGRIS Baptist Medical Center, Oklahoma City, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LVAD Recipients
Started | 211
Completed | 211
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LVAD Recipients
Number analyzed (Participants) | 211
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 211
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 163
Region of Enrollment [Number; unit: participants]
  United States | 211

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Left Ventricular Recovery and LVAD Explant
Description: Noninvasive determination of left ventricular function using novel echocardiographic imaging methods and routine clinical assessments to optimize markers of left ventricular recovery. These markers would determine LVAD patients with cardiac recovery who no longer needed LVAD support.
Time Frame: Number of participants who had LV recovery and LVAD explant over 3 years.
Population: The outcome measured were the number of patients who had cardiac recovery and who no longer required LVAD support and had successful LVAD explant. Of 211 LVAD recipients, there were 8 who had successful LVAD explant
Measure: Count of Participants; unit: Participants
Arm/Group | LVAD Recipients
Number analyzed (Participants) | 211
Participants | 8

2. Secondary Outcome: Refine and Test Feedback Control Algorithm That Allows Precise Prescription of Cardiac Loading Through Synchronized and Asynchronized LVAD Operation With Native Left Ventricular Contraction
Time Frame: Measured at Year 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | LVAD Recipients
Serious Adverse Events (participants affected / at risk) | 0/211
Other Adverse Events (participants affected / at risk) | 0/211

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes